CLINICAL TRIAL: NCT00595270
Title: Long Term Persistence and Effect of a Booster Dose of the Japanese Encephalitis Vaccine IC51
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IC51-305
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Results first posted 2014-03-07 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-02

CONDITIONS: Japanese Encephalitis
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IC51 (Other): In study IC51-305, subjects who had received IC51 in study IC51-304 were tested for seroconversion 6 months after the first vaccination. Subjects who had protective titers were again tested for persistence of immunity at 12 months after the first immunization,whereas subjects who had titers below the seroconversion threshold by Month 6 received a booster dose of 1x6 mcg IC51 at Month 11. Their immune response was also assessed at Month 12. Thereafter, subjects who had no protective titer by Month 12 received a booster dose of 1x6 mcg IC51 at Month 23, regardless of prior treatment; and neutralizing antibody titers were reassessed at Month 24. Subjects who had protective titers at month 12 did not receive a booster at Month 23, and their neutralizing antibody titer was also assessed at Month 24.
  Interventions: Biological: IC51

INTERVENTIONS:
Biological: IC51
  Other Names: Japanese Encephalitis purified inactivated vaccine

SUMMARY:
The study investigates the long term persistence the Japanese encephalitis vaccine IC51 and the need of a booster dose

DETAILED DESCRIPTION:
This is an open label, non-randomized multi-center phase 3 follow-up study. All volunteers having completed trial IC51-304 (NCT00595790) will be enrolled into this trial at 2 sites

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Written informed consent obtained prior to study entry
* Subjects correctly included in and having completed study IC51-304 according to the protocol.

Exclusion Criteria:

* Use of any other investigational or non-registered drug or vaccine in addition to the study vaccine during the study period
* Immunodeficiency including post-organ-transplantation or immunosuppressive therapy
* Pregnancy, lactation or unreliable contraception in female subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2005-10; Primary Completion 2007-09 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Eder, Study Director — Valneva Austria GmbH

RESULTS

PARTICIPANT FLOW:
Groups:
- IC51 2 x 6 µg; IC51 1 x 12 µg; IC51 1 x 6 µg: treatment group in preceeding study IC51-304
Period: Overall Study
Arm/Group | IC51 2 x 6 µg | IC51 1 x 12 µg | IC51 1 x 6 µg
Started | 116 | 117 | 116
Completed | 110 | 107 | 108
Not Completed | 6 | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IC51 2 x 6 µg | IC51 1 x 12 µg | IC51 1 x 6 µg | Total
Number analyzed (Participants) | 116 | 117 | 116 | 349
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 109 | 108 | 106 | 323
  >=65 years | 7 | 9 | 10 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 60 | 57 | 184
  Male | 49 | 57 | 59 | 165
Region of Enrollment [Number; unit: participants]
  Europe | 116 | 117 | 116 | 349

OUTCOME MEASURES:

1. Primary Outcome: Long Term Immunogenicity of IC51 Vaccine 24 Months After the Primary Vaccination
Description: Seroprotection rate (SPR) (anti-JEV neutralizing antibody titer ≥ 1:10) 24 months (M24) after the primary vaccination - imputed; Persistence of immunogenicity (SPR) at M24 defined as:
  * pos. (positive) (persistent): Subjects
    * with a non-missing, pos. seroconversion at D56 (Study IC51-304) and
    * without booster at M11 or M23 and
    * with non-missing, seroprotection (SP) pos. PRNT50 at M6 or M12 and
    * with non-missing, SP pos. PRNT50 at M24
  * neg. (negative) (non-persistent): Subjects with
    * missing or neg. seroconversion at D56 (Study IC51-304) or
    * booster at M11 or at M23, or
    * non-missing, SP neg. PRNT50 at M6 or M12 or
    * missing PRNT50 at both M6 and M12 or
    * missing or SP neg. PRNT50 (serum dilution giving 50% reduction in plaques in a Plaque Reduction Neutralization Test) at M24
Time Frame: - 24 months
Population: ITT (Intent-To-Treat) Population: included all subjects rolled over from study IC51-304; analyzed according to treatment to which they were randomized in IC51-304
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IC51 2 x 6 µg | IC51 1 x 12 µg | IC51 1 x 6 µg
Number analyzed (Participants) | 116 | 117 | 116
percentage of participants | 56 [39.4 to 57.3] | 7 [3.0 to 11.9] | 5 [1.8 to 9.6]

2. Secondary Outcome: SPR 24 Months After the Primary Vaccination (Observed)
Description: Persistence of immunogenicity (SPR) at M24 (observed) defined as :
  * positive (persistent): Subjects
    * with a non-missing, positive seroconversion at D56 (Study IC51-304), and
    * who did not receive a booster dose at Visit 2 (M11) or Visit 4 (M23), and
    * with a non-missing, SP positive PRNT50 result at Visit 1 (M6) or Visit 3 (M12), and
    * with a non-missing, SP positive PRNT50 result at Visit 5 (M24)
  * negative (non-persistent): Subjects
    * with missing or negative seroconversion at D56 (Study IC51-304), or
    * who did receive a booster dose at Visit 2 (M11) or at Visit 4 (M23), or
    * with a non-missing, SP negative PRNT50 result at Visit 1 (M6) or Visit 3 (M12), or
    * with a missing PRNT50 result at both Visit 1 (M6) and Visit 3 (M12), or
    * with a non-missing, SP negative PRNT50 result at Visit 5 (M24)
Time Frame: 24 months
Reporting Status: Not Posted

3. Secondary Outcome: Persistent and Actual SPR 6, 12 and 24 Months After Primary Vaccination
Time Frame: - 24 months
Reporting Status: Not Posted

4. Secondary Outcome: Persistent and Actual GMT 6, 12 and 24 Months After Primary Vaccination
Time Frame: 24 months
Reporting Status: Not Posted

5. Secondary Outcome: SCR 1 Month After the Booster Doses
Time Frame: 1 month
Reporting Status: Not Posted

6. Secondary Outcome: GMT 1month After Booster Doses
Time Frame: 1 month
Reporting Status: Not Posted

7. Secondary Outcome: Safety Profile of IC51
Time Frame: study duration
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | IC51 2 x 6 µg | IC51 1 x 12 µg | IC51 1 x 6 µg
Serious Adverse Events (participants affected / at risk) | 4/116 | 4/117 | 3/116
Other Adverse Events (participants affected / at risk) | 61/116 | 69/117 | 64/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IC51 2 x 6 µg (N=116) | IC51 1 x 12 µg (N=117) | IC51 1 x 6 µg (N=116)
Appendicitis (Infections and infestations) | 1 | 0 | 0
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 1 | 0 | 0
Uterine Prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Paranasal Sinus Discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hysterectomy (Surgical and medical procedures) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IC51 2 x 6 µg (N=116) | IC51 1 x 12 µg (N=117) | IC51 1 x 6 µg (N=116)
Fatique (General disorders) | 5 | 7 | 6
Influenza Like Ilness (General disorders) | 7 | 5 | 6
Nasopharyngitis (Infections and infestations) | 12 | 13 | 11
Headache (Nervous system disorders) | 10 | 12 | 13
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 0
Nausea (Gastrointestinal disorders) | 1 | 6 | 4
Toothache (Gastrointestinal disorders) | 2 | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1
Sinusitis (Infections and infestations) | 3 | 0 | 1
Accidental Poisoning (Injury, poisoning and procedural complications) | 1 | 3 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 5
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 2
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 4
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 2 | 0
Induration (General disorders) | 1 | 0 | 2
Injection Site Pain (General disorders) | 0 | 2 | 1
Herpes Zoster (Infections and infestations) | 1 | 0 | 2
Lower Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 2
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 2 | 0
Haematocrit Decreased (Investigations) | 0 | 2 | 0
Haemoglobin Decreased (Investigations) | 0 | 2 | 0
Red Blood Cell Count Decreased (Investigations) | 0 | 2 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other